CLINICAL TRIAL: NCT01173926
Title: A Trial Comparing the Pharmacokinetic and Pharmacodynamic Properties Between NN5401 and NN1250 and Between NN5401 and Insulin Aspart in Subjects With Type 1 Diabetes
Brief Title: Comparison of the Effect of NN5401 With the Effect of NN1250 and Insulin Aspart in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-3857; U1111-1114-9348 (Other: WHO); 2010-019641-26 (EudraCT Number)
Record Dates: First submitted 2010-07-30; First posted 2010-08-02 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; insulin degludec, insulin aspart drug combination; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IAsp (Experimental)
  Interventions: Drug: insulin aspart
- IDeg (Experimental)
  Interventions: Drug: insulin degludec
- IDegAsp (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart

INTERVENTIONS:
Drug: insulin degludec — Each trial participant will receive one single dose of each trial product in varying order (NN5401, NN1250 and insulin aspart) on 3 separate dosing visits. The trial products will be administered subcutaneously (under the skin).
  Arms: IDeg
Drug: insulin degludec/insulin aspart — Each trial participant will receive one single dose of each trial product in varying order (NN5401, NN1250 and insulin aspart) on 3 separate dosing visits. The trial products will be administered subcutaneously (under the skin).
  Arms: IDegAsp
Drug: insulin aspart — Each trial participant will receive one single dose of each trial product in varying order (NN5401, NN1250 and insulin aspart) on 3 separate dosing visits. The trial products will be administered subcutaneously (under the skin).
  Arms: IAsp

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare the blood glucose-lowering effect of NN5401 (insulin degludec/insulin aspart, IDegAsp) with NN1250 (insulin degludec, IDeg) and insulin aspart (IAsp) in subjects with type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months.
* Body mass index 18.0-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day).
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve | From 0 to 6 hours after single-dose (only for IDeg and IDegAsp)
Area under the glucose infusion rate curve | From 6 to 24 hours after single-dose (only for IDegAsp and IAsp)

SECONDARY OUTCOMES:
Area under the serum insulin degludec concentration-time curve | From 0 to 120 hours after single-dose (only for IDeg and IDegAsp)
Area under the serum insulin aspart concentration-time curve | From 0 to 12 hours after single-dose (only for IDegAsp and IAsp)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com